CLINICAL TRIAL: NCT06133803
Title: Lovenox With Aspirin in Thawed Blastocyst Transfer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fertility Center of Las Vegas (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FCLV 2023-2
Record Dates: First submitted 2023-11-10; First posted 2023-11-18 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-11

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Enoxaparin; Aspirin; Embryo Transfer

STUDY DESIGN:
Intervention Model Description: Randomized trial comparing treatment to controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Patients randomized to receive aspirin and Lovenox will begin taking one "low dose" 81mg aspirin and one 40mg injection of Lovenox daily, on the day of progesterone start.
  Interventions: Drug: Lovenox; Drug: Aspirin; Procedure: Embryo transfer
- Control Arm (Active Comparator): This arm receives neither medication.
  Interventions: Procedure: Embryo transfer

INTERVENTIONS:
Drug: Lovenox — A low-molecular-weight heparin, 40mg daily injection.
  Arms: Treatment Arm
Drug: Aspirin — Aspirin 81mg daily tablet.
  Arms: Treatment Arm
Procedure: Embryo transfer — Embryo transfer

SUMMARY:
This prospective randomized trial will compare outcomes in patients receiving aspirin in combination with a low-molecular weight heparin and those under this center's standard protocol receiving neither medication, in order to determine if these medications may improve success rates.

DETAILED DESCRIPTION:
This prospective randomized trial will compare outcomes in patients receiving aspirin (81mg daily) in combination with a low-molecular weight heparin (LMWH) (enoxaparin (Lovenox®), 40mg daily subcutaneous injection) and those under this center's standard protocol receiving neither medication, in order to determine if these medications may improve success rates.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient 18-42 years of age with frozen embryos or oocytes seeking embryo transfer.
2. Use of pre-implantation genetically tested (PGT) blastocysts is allowed but not required.
3. Use of donated embryos or embryos derived from donated eggs is allowed.
4. Prior history of successful, failed, and/or canceled IVF cycles are allowed.

Exclusion Criteria:

1. Minor (age<18 years).
2. Currently pregnant.
3. Unable to provide informed consent in English.
4. Gestational carrier or "surrogate".
5. Blastocysts frozen at another center (Oocytes frozen elsewhere is acceptable).
6. Subject intending or having "natural cycle" thaw transfer with an active ovarian follicle present.
7. Currently participating in any other research study.
8. Subject already had an embryo transfer under this study.
9. History of thrombocytopenia (reduced platelets), bleeding disorders, or routinely using anti-coagulant medication.
10. Hypersensitivity to aspirin, heparin, or benzyl alcohol.
11. Anyone for whom the physician assesses this protocol is inappropriate or unsafe.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female seeking pregnancy.
Enrollment: 130 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Serum hCG level | 5 days post transfer
  Serum hCG level

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Shapiro, MD, PhD, Principal Investigator — Fertility Center of Las Vegas
Locations (1):
- Fertility center of Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No